CLINICAL TRIAL: NCT05135247
Title: Cardiac Autonomic Modulation in Older Hypertensive Individuals Submitted to Different Types of Physical Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nereida Kilza da Costa Lima, Associated Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.092.824
Record Dates: First submitted 2021-11-09; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Autonomic Dysfunction
Keywords: older individuals; heart rate variability; physical training; hypertension
MeSH Terms: conditions — Primary Dysautonomias; Hypertension | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The individuals were randomized into four groups: continuous aerobic training (CA), interval aerobic training (IA), resistance training (R), and control (C), which performed physical exercises three times a week for twelve weeks, with a total of 36 sessions. The tilt test was performed before and after the research protocol. Individuals in the control group were only encouraged to maintain their usual activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- continuous aerobic training (CA) (Experimental): The CA group was trained with 70% of maximum heart rate (MHR) for 30 minutes.
  Interventions: Other: Exercise
- resistance training (R) (Experimental): The R sessions consisted of a set of each proposed exercise: sitting bench press, legpress, back row, leg extension, shoulders high pull, seated leg curl, biceps curls, standing calf, triceps in the pulley, and abdominal crunches, with 8 - 10 repetitions with 75% 1MR.
  Interventions: Other: Exercise
- interval aerobic training (IA) (Experimental): The IA group was submitted to exercise intensities of 60% for 2 minutes and 80% for 2 minutes, alternately, with a total of 30 minutes.
  Interventions: Other: Exercise
- control (C) (No Intervention): Individuals in the control group maintained their usual activities.

INTERVENTIONS:
Other: Exercise — 3 different types of training or control
  Arms: continuous aerobic training (CA); interval aerobic training (IA); resistance training (R)

SUMMARY:
Sixty-one sedentary older hypertensive individuals were randomized to four groups: continuous aerobic training (CA), interval aerobic training (IA), resistance training (R), and control (C) group. The protocol included 3 sessions of training by week for 12 weeks. C individuals were instructed to continue their usual activities. They were submitted to the passive tilt test before and after the research protocol, evaluating the heart rate (HR), low frequency (LF) and high frequency (HF) bands, detrended fluctuation analysis (DFAα1) and entropy

DETAILED DESCRIPTION:
The individuals were randomized into four groups: continuous aerobic training (CA), interval aerobic training (IA), resistance training (R), and control (C), which performed physical exercises three times a week for twelve weeks, with a total of 36 sessions. The tilt test was performed before and after the research protocol. Individuals in the control group were only encouraged to maintain their usual activities.

For the analysis of HRV, the baseline conditions (resting in the supine position) were determined, followed by the passive postural maneuver, which characterizes the tilt test (table til tat 70 °) in order to determine the following variables:

* HR: heart rate (sympathetic action)
* LF: Low frequency band (Modulated predominantly by the sympathetic system)
* HF: High frequency band (Modulated predominantly by the parasympathetic system)
* Entropy: data complexity or irregularity index showing that, the higher the values, the better the HRV.
* DFAα1 (short term detrended fluctuation analysis)

ELIGIBILITY:
Inclusion Criteria:men and women 60-year-old or older, extensively using prescription antihypertensive drugs, and having no previous experience with physical training -

Exclusion Criteria:

* • Positive treadmill test (TT) for ischemia

  * Related left ventricular systolic dysfunction of any degree
  * Presence of arrhythmias
  * Use of β-blockers
  * Use more than seven doses of ethyl alcohol per week
  * Renal insufficiency
  * Diabetes
  * Hyper- or hypothyroidism
  * Limiting lung disease
  * Osteomioarticular impairment that would limit exercise performance
  * SBP ≥160 and/or DBP ≥ 100 mmHg on baseline

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Heart rate | 12 weeks
  Heart rate was obtained before and after the protocol by electrocardiogram, performed before and after tilt test at each time.
Low frequency band | 12 weeks
  Low frequency band was obtained before and after the protocol by electrocardiogram, performed before and after tilt test at each time.The electrical signal from the electrocardiogram was filtered and amplified. The amplified signals were processed by ananalog-digital converter (DI-720, DATAQ Instruments, Akron, OH, USA) and sampled (1000 hz per channel) by a computer program (Windaq, DATAQ, Akron, OH, USA) installed in an IBM/PC computer.
High frequency band | 12 weeks
  High frequency band was obtained before and after the protocol by electrocardiogram, performed before and after tilt test at each time.The electrical signal from the electrocardiogram was filtered and amplified. The amplified signals were processed by ananalog-digital converter (DI-720, DATAQ Instruments, Akron, OH, USA) and sampled (1000 hz per channel) by a computer program (Windaq, DATAQ, Akron, OH, USA) installed in an IBM/PC computer.
Entropy | 12 weeks
  Entropy was obtained before and after the protocol by electrocardiogram, performed before and after tilt test at each time.The electrical signal from the electrocardiogram was filtered and amplified. The amplified signals were processed by ananalog-digital converter (DI-720, DATAQ Instruments, Akron, OH, USA) and sampled (1000 hz per channel) by a computer program (Windaq, DATAQ, Akron, OH, USA) installed in an IBM/PC computer.
Short term detrended fluctuation analysis | 12 weeks
  Short term detrended fluctuation analysis obtained before and after the protocol by electrocardiogram, performed before and after tilt test at each time.The electrical signal from the electrocardiogram was filtered and amplified. The amplified signals were processed by ananalog-digital converter (DI-720, DATAQ Instruments, Akron, OH, USA) and sampled (1000 hz per channel) by a computer program (Windaq, DATAQ, Akron, OH, USA) installed in an IBM/PC computer.

IPD SHARING:
Plan to Share IPD: Yes
Individual data of volunteers, without identification, can be provided if requested by other authors, through contact with the main researcher
Supporting Information: Study Protocol
Time Frame: Data will be made available after the publication of the study, with no time to end sharing
Access Criteria: contact with the main researcher